CLINICAL TRIAL: NCT00530660
Title: An Open-label Phase II Study to Assess the Immunogenicity and Safety of a Booster Vaccination With a Heterologous Vero Cell-Derived Whole Virus H5N1 Influenza Vaccine in a Healthy Young Adult Population (Follow Up to Study 810501)
Brief Title: Safety and Immunogenicity Study of a Booster Vaccination With a Non-Adjuvanted H5N1 Influenza Vaccine (Follow Up to Study 810501)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alachua Government Services, Inc. (Industry)
Responsible Party: Simone Deutschel, Clinical Project Manager, Baxter Healthcare Corporation
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 810703
Record Dates: First submitted 2007-09-14; First posted 2007-09-17 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2008-12

CONDITIONS: Influenza
Keywords: Pandemic influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: H5N1 influenza vaccine (whole virion, Vero cell-derived), 7.5 µg HA antigen, non-adjuvanted — All subjects who have completed the Day 42 visit at the Austrian study site in Study 810501 will be invited to receive a booster vaccination, 12 to 17 months after the first vaccination with the A/Vietnam/1203/2004 influenza vaccine administered in Study 810501, with a heterologous whole virion, Vero cell-derived influenza vaccine containing 7.5 mg A/H5N1/Indonesia/05/2005 hemagglutinin (HA) antigen in a non-adjuvanted formulation.

SUMMARY:
The purpose of this Phase II follow-up study (to study 810501) is to assess the immunogenicity and safety of a booster vaccination with a non-adjuvanted H5N1 influenza vaccine administered 12 to 17 months after a two-dose regimen of different doses of an adjuvanted or non-adjuvanted H5N1 influenza vaccine in a healthy young adult population. A data safety monitoring board will review the safety data after the booster vaccination. The H5N1 influenza antibody persistence 180 days after the booster vaccination will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

Subjects who participated in Study 810501 will be eligible for participation in the study if they:

* Completed the Day 42 visit in study 810501
* Have an understanding of the study, agree to its provisions, and give written informed consent prior to study entry
* Are clinically healthy, as determined by the Investigator's clinical judgment through collection of medical history and performance of a physical examination
* Agree to keep a daily record of symptoms for the duration of the study
* If female and capable of bearing children, have a negative urine pregnancy test result at study entry and agree to employ adequate birth control measures for the duration of the study

Exclusion Criteria:

* Have a history of vaccination with an H5N1 influenza virus since the second vaccination in study 810501
* Have had an allergic reaction to one of the components of the vaccine since the second vaccination in Study 810501
* Have been diagnosed with a significant neurological, cardiovascular, pulmonary (including asthma), hepatic, rheumatic, autoimmune, hematological, renal or metabolic disorder since the second vaccination in Study 810501
* Are unable to lead an independent life as a result of either physical or mental handicap
* Suffer from any kind of immunodeficiency since the second vaccination in Study 810501
* Suffer from a disease or were undergoing a treatment within 30 days prior to the scheduled booster vaccination or are currently undergoing a form of treatment that can be expected to influence immune response. Such treatment includes, but is not limited to, systemic or high dose inhaled (>800µg/day of beclomethasone dipropionate or equivalent) corticosteroids, radiation treatment or other immunosuppressive or cytotoxic drugs
* Have had severe allergic reactions or anaphylaxis since the second vaccination in Study 810501
* Have a rash, dermatologic condition or tattoos which may interfere with injection site reaction rating
* Have undergone systemic corticoid therapy within 30 days prior to study entry
* Have a functional or surgical asplenia
* Have a known or suspected problem with alcohol or drug abuse
* Were administered an investigational drug within six weeks prior to study entry or are concurrently participating in a clinical study that includes the administration of an investigational product
* Are a member of the team conducting this study or are in a dependent relationship with the study investigator. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the investigator If female, are pregnant or lactating

Ages: 18 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Estimated)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects with antibody response to the vaccine strain (A/Indonesia/05/2005) associated with protection 21 days after the booster vaccination (HI antibody titer >= 1:40 or MN titer >= 1:20) | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Baxter BioScience Investigator, Principal Investigator — Baxter Healthcare Corporation
Locations (1):
- University Hospital, Department of Clinical Pharmacology, General Hospital Vienna, Vienna, Austria

REFERENCES:
- [Derived] Ehrlich HJ, Muller M, Fritsch S, Zeitlinger M, Berezuk G, Low-Baselli A, van der Velden MV, Pollabauer EM, Maritsch F, Pavlova BG, Tambyah PA, Oh HM, Montomoli E, Kistner O, Noel Barrett P. A cell culture (Vero)-derived H5N1 whole-virus vaccine induces cross-reactive memory responses. J Infect Dis. 2009 Oct 1;200(7):1113-8. doi: 10.1086/605608. PMID 19712040